CLINICAL TRIAL: NCT07041229
Title: The First Prospective Randomized Study of the Removal of Large Benign Epithelial Neoplasms of the Colon by the EMR and ESD Method in Moscow, Russia.
Brief Title: Comparison of Methods for Removing Large Benign Broad-based Epithelial Neoplasms of the Colon: ESD and EMR.
Acronym: ESDEMR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06111985_01; 1503-6/23 (Other: Moscow Center for Innovative Technologies in Healthcare)
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2024-12

CONDITIONS: Benign Colon Tumors
Keywords: ESD, EMR
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMR (Experimental): The time of removal, the number of fragments, complications, its immediate and remote results are assessed,histology result
  Interventions: Procedure: EMR; Procedure: ESD
- ESD (Experimental): . The time of removal, the number of fragments, submucous fibrosis and its degree, complications, and immediate and long-term results are assessed,histology result
  Interventions: Procedure: EMR; Procedure: ESD

INTERVENTIONS:
Procedure: EMR — 3-4 ml of high-osmolar solution or saline solution stained with indigo carmine are introduced into the submucosal layer under the formation. The formation and the surrounding mucous membrane (at least 5 mm from the edge of the formation) are removed using a standard diathermic polypectomy loop available to the operator. The formation is removed using electric current in the EndocatQ mode. After the formation is removed, the resection site is examined in white light, then virtual chromoscopy (NBI), and then examined with magnification. If residual tissue of the formation is detected, it is removed using the same technique. If the removal of residual tissue of the formation was performed by another method, indicate which one and why.
  The removed formation is extracted using a snare loop; if it is removed in parts, then all fragments, if possible, are extracted through the aspiration channel of the endoscope; for large fragments, a snare loop is used.
  Other Names: Endoscopic mucosal resection
Procedure: ESD — After assessing the boundaries of the formation, a mark is made at least 5 mm from the edge, then a circular or semicircular incision of the mucosa is made, after which the formation is removed by dissection of the submucosal layer using a scarecrow knife, a knife with a ceramic head at the end in EndocutQ mode, spray-coag swift-coag. The EDPS technique - a tunnel method, will also be used where feasible. The essence of the technique is a semilunar incision of the mucous membrane, retreating from the marks, and creating a tunnel under the formation to the proximal edge of the marks, with subsequent cutting off of the formation along the edges. The removed neoplasm is extracted and stretched on a plate. After removal, the edges and bottom of the wound are assessed, if necessary, prophylactic coagulation of visible vessels and clipping are performed.
  Other Names: Endoscopic submucosal dissection

SUMMARY:
Benign epithelial neoplasms of the colon are a significant problem of colorectal surgery and health care not only because of their malignant potential, but also because of their prevalence among the working-age population. Adenomas are more often detected in men than in women (OR = 1.77; 95% CI = 1.66-1.89), increasing in men from 25% at 50-54 years to 39% in people over 70 years old and in women from 15% at 50-54 years to 26% at 70 years of age (p < 0.001) [1]. Colonoscopy is the gold standard among all methods for diagnosing adenomas and adenocarcinomas of the colon. Endoscopic removal of colorectal polyps reduces the incidence and mortality from colorectal cancer (CRC) and is considered a necessary skill for all endoscopists performing colonoscopy [2, 6]. Endoscopic mucosal resection (EMR) was developed in 1984 by M. Tada et al. as a new technique for removing epithelial lesions of the gastrointestinal tract [181]. There are a number of aspects that cause additional complications during mucosectomy, such as convergence of folds, localization of large polyps between two folds, tumor spread beyond two folds, which are factors in tumor fragmentation and require additional study of their impact on long-term treatment outcomes. It is important to note that removal of colon tumors by fragmentation technique is associated with increased recurrence rate, however, in most cases these recurrent lesions are small in size and can be easily removed during dynamic colonoscopy. Predictably high recurrence rate during tumor fragmentation during removal indicates non-radical nature of the intervention performed and safety of this manipulation should be proven. Endoscopic submucosal dissection (ESD) is a relatively new method for removing superficial gastrointestinal neoplasms and was described at the end of the 20th century [85]. The development of the submucosal dissection technique was motivated by the difficulty of removing formations larger than 20 mm in a single block by endoscopic resection of the mucosa. Also, the association of tumor fragmentation during resection with a high risk of local recurrence and the difficulty of morphological evaluation of the removed specimen [133, 136, 190]. However, endoscopic submucosal dissection is a lengthy and energy-consuming procedure. According to Japanese authors, the average time for endoscopic submucosal dissection is 48.5-60 min. [77, 89], and, according to European scientists, the time for performing such interventions ranges from 142 to 176 minutes [7, 78, 144, 187]. According to Japanese clinical guidelines, the preferred method for removing large epithelial neoplasms of the colon with suspected intramucosal invasion is ESD, and European and American guidelines talk about the possible use of EMR, including in parts. In addition, unlike Japanese guidelines, where it is considered unsafe to remove a neoplasm in parts in assessing its radicality, Western guidelines allow the use of EMR in parts. Thus, endoscopic resection of the mucous membrane and endoscopic dissection in the submucosal layer are currently successfully used in the treatment of epithelial formations, but the advantages and disadvantages of each technique for a particular type of neoplasm, its histological nature and localization require systematization and clarification. The place of endoscopic mucosal resection and submucosal dissection in the removal of epithelial lesions of the colon has not been definitively established. Technical aspects, risk factors for complications, and long-term results of these types of endoscopic interventions require additional analysis.

Endoscopic interventions on the colon are accompanied by a certain percentage of complications. The most common complications of endoscopic removal of colon neoplasms are bleeding and perforation, the frequency of which varies from 0.08% to 10% depending on the analyzed method and patient sample [93, 120]. Given the wide variability of the available data, the influence of various factors on the frequency of complications requires additional study due to the need to identify correctable variables.

In June 2022, a group of authors proposed to the world community of specialists a new classification of complications in endoluminal endoscopy of the gastrointestinal tract for standardized assessment and analysis of the safety of endoscopic interventions [1] - "AGREE" (acronym for Adverse events GastRointEstinal Endoscopy) The authors of the classification also recommend recording any complications that arise, both at the stage of preparation for the planned endoscopic intervention (regardless of whether it was ultimately performed or not), and in those30 days after the intervention.[1]. It is these provisions of the AGREE classification that remain controversial and require more careful discussion [3]. In any case, in our opinion, at least a cause-and-effect relationship should be established between the action and the complication.

DETAILED DESCRIPTION:
Objective of the study: to prospectively compare the immediate, immediate and remote results of endoscopic mucosal resection through an endoscope and endoscopic submucosal dissection performed for non-invasive large-sized (20 mm or more) broad-based epithelial lesions of the colon.

Study objectives:

1. To evaluate the accuracy of ultra-high-resolution colonoscopy in white, ultra-clear and narrow-spectrum light with magnification in predicting the histological structure and risks of invasion of large-sized broad-based epithelial lesions of the colon.
2. To conduct a comparative assessment of the accuracy of angio-CT/MRI, probe EUS and second-generation narrow-band endoscopy with magnification in determining the depth of invasion and the probability of lymphoregional metastasis of superficial epithelial neoplasms of the colon with malignancy.
3. To evaluate the effectiveness of endoscopic ultrasound in predicting submucosal fibrosis and its impact on surgical treatment tactics, and to compare the obtained data with the intraoperative picture using the fibrosis classification scale.
4. To conduct a comparative assessment of the completeness (in one block/in parts; R0/R1) and depth of resection of large-sized epithelial lesions of the colon on a broad base according to endoscopic and morphological criteria in EMR and ESD.
5. To study the immediate results of EMR and ESD, including conversion and intervention refusal factors.
6. To determine the risk factors for recurrence after endoscopic removal of large epithelial neoplasms of the colon and to develop an algorithm for their diagnosis and prevention
7. To assess possible intra- and postoperative complications during endoscopic removal of large epithelial neoplasms (bleeding, perforation, postcoagulation syndrome) of the colon using the AGREE endoscopic complication scale and to develop methods for their prevention and treatment.
8. To assess the effectiveness of the RDI regimen both for the prevention of an intraoperative source of bleeding and for detecting a source of bleeding during EMR/ESD
9. To study comparative indicators of the number of tumor recurrences in the immediate and late periods after endoscopic intervention (from 6 months to 5 years), and the effect of the EMR method and additional ablation of the edges of the wound bottom on the incidence of recurrent formations

General characteristics of the clinical study. Design: prospective, randomized, controlled study. It is planned to include at least 110 patients in the study until statistically reliable indicators are obtained for all analyzed parameters, who will undergo EMR or ESD for large-sized (20-60mm) non-invasive epithelial formations of the colon on a broad base. The method of choosing the operation will be determined using a random number generator (randomizer).

Patient inclusion criteria:

1. Patient with benign non-invasive epithelial formations of the colon on a broad base (Is and II types), 20-60mm in size
2. Age ≥ 18 years.
3. Signed informed voluntary consent for colonoscopy and removal of formations using the studied methods.

Patient exclusion criteria:

1. More than one large epithelial formation on a broad base
2. Colon formations less than 20 and more than 60 mm
3. Recurrent nature of the formation.
4. Reasonable suspicion of the presence of an invasive formation (cancer), including with invasion into the submucosal layer based on the results of preoperative assessment (NICE - 3; JNET - 3; Kudo - Vn).
5. The presence of a widespread malignant tumor in any part of the colon.
6. Use of other methods of endoscopic removal of the formation.
7. IBD.
8. Infectious disease requiring systemic therapy
9. Patient on hemodialysis
10. Uncorrectable coagulopathy (INR> 1.5), inability to discontinue antithrombotic drugs.
11. Refusal to participate in the study.
12. General contraindications to endoscopic examination.

All patients were randomly divided into 2 main groups (using a randomizer) using block stratification randomization: EMR Group and ESD Group.

https://randomus.ru/quick?from=1&to=110&count=55&norepeat=1&sort=1

ESD (55) patients with numbers:

5, 6, 7, 9, 13, 16, 17, 18, 19, 22, 24, 25, 28, 29, 30, 32, 33, 35, 36, 37, 38, 40, 42, 44, 47, 49, 50, 51, 58, 59, 62, 64, 65, 69, 70, 74, 75, 76, 77, 78, 79, 81, 85, 89, 93, 94, 95, 96, 98, 99, 103, 105, 106, 108, 110

Other patients - EMR (55):

1,2,3,4,8,10,11,12,14,20,21,23,26,27,31,34,39,41,43,45,46,48,52,53,54,55,56,57,60,61,63,66,67,68,71,72,73,80,83,84,86,87,88,90,91,92,97,100,101,102,104, 109 In the EMR group, it is planned to additionally divide patients into 2 main groups (using a randomizer) using block stratification randomization: EMR Group and EMR + Group ablation.

https://randomus.ru/quick?from=1&to=56&count=28&norepeat=1&sort=1

EMR +APC (28 patients): 2, 5, 6, 7, 11, 12, 18, 19, 22, 24, 26, 28, 30, 32, 34, 35, 37, 38, 39, 41, 42, 43, 44, 45, 46, 47, 50, 51 The rest are EMR (28 patients)

It is planned to evaluate the following patient characteristics:

1. Gender.
2. Age.
3. Taking aspirin (or analogs) and/or indirect anticoagulants
4. The degree of concomitant pathology, expressed in the concept of surgical-anesthesiological risk according to the ASA scale.
5. History of abdominal surgery
6. History of inflammatory diseases of the abdominal organs, including diverticulitis, usually leading to the formation of adhesions involving the colon,

The following characteristics of the study are planned to be assessed:

1. Nature of preparation (compliance/non-compliance with the recommended diet; drug(s) used, split preparation or not, time from the last dose to the start of colonoscopy), quality of preparation (according to the Boston scale).
2. Presence of sedation (Yes/No).
3. Use of a distal cap (Yes/No).

The following endoscopic characteristics of the epithelial formation are planned to be assessed:

1. Localization (according to anatomical landmarks), preferably indicating the number of haustra from significant landmarks; as well as on the fold, through the fold in the interfold space.
2. Size of the formation (mm) using a ruler;
3. Type according to the Paris Classification of Epithelial Neoplasia and the Classification of Laterally Spreading Tumors;
4. Assessment of the surface microstructure according to NICE, JNET, WASP, Kudo.
5. Assessment of invasion and submucosal fibrosis using EUS probes

The following characteristics of EMR and ESD are planned to be assessed:

1. Method of removal (EMR with injection of a high-osmolar solution (gelofusin) into the submucosal layer or ESD);
2. Removal time (from the moment the loop is brought into the field of view until complete removal of the formation or from the beginning of the incision);
3. Method of removal (in fragments or as a single block, ESD or combined ESD, or impossibility of removal);
4. Completeness of removal according to high-resolution endoscopy, virtual chromoscopy and magnification at the end of the intervention (within healthy tissue/no), which will be confirmed by taking a biopsy (4 fragments) from the edges of the resection wound after EMR
5. Evaluate the EUS data with intraoperative data and pathomorphological conclusion data regarding the presence of fibrosis and neoplasm invasion.
6. Removal of the specimen (removed/lost) and the reason for loss.
7. Use of prophylactic clipping (Yes/No) and indications for its use: deep post-resection defect (up to and including the muscular layer); intestinal perforation; inability to achieve hemostasis; for social reasons (doctor, relatives...)
8. After performing EMR, use a randomizer to select a method for preventing recurrence of the formation in the group - ablation with the tip of the loop and a control group where ablation will not be performed
9. Type and nature of adverse events according to the AGREE scale
10. In case of damage to the wall of the colon, it will be assessed according to the scale of damage to the wall of the colon and, depending on this, the treatment tactics will be selected.

It is planned to evaluate the following characteristics in the postoperative period:

1. The presence of abdominal pain syndrome (Yes/No)
2. Temperature Yes/No (within 24 hours, above 37.2).
3. Type, time of occurrence and nature of adverse events (bleeding, perforation, postcoagulation syndrome).
4. Type of observation after removal (outpatient/inpatient). If inpatient, for how long.
5. Compliance with a diet in the postoperative period (yes/no).
6. Use of antibiotics (yes/no).
7. Use of hemostatics (yes/no).
8. If postcoagulation syndrome is suspected - assessment of C reactive protein, assessment of leukocytes in the blood

It is planned to assess the following morphological characteristics of the formation:

1. Fragmentation of the formation (yes/no)
2. Histological structure of the formation (examination of the removed specimen, according to the WHO and Vienna classification).
3. Morphological assessment of the completeness of removal (assessment of the specimen) - R0 - no cells of the formation along the resection line, R1 - there are cells of the formation along the resection line, Rx - the formation is removed in fragments or the status of the resection boundaries cannot be determined.
4. Morphological assessment of the edges of the p/o wound after EMR - 4 tissue fragments - one from each edge

Technique of endoscopic intervention. To prepare for colonoscopy, it is recommended to: adhere to a low-residue diet for 2 days (the 3rd and 2nd day before the endoscopic intervention); drink only clear liquids the day before; use full-volume PEG-based drugs (Fortrans) or a low-volume sulfate-based drug (Eziclen) in split mode.

After visualization of the formation, its localization is assessed, its type according to the Paris classification of epithelial neoplasia, its size compared to the diameter of the catheter ("shirt") of the loop and the polypectomy loop itself in the open state. (If technically possible, welcome(the use of an endoscopic ruler is required). The nature of the surface of the formation is assessed in white light, in TXI mode, and using virtual chromoscopy according to NICE, WASP; with magnification - according to JNET and, if necessary, according to Kudo with a 0.5-1.0% indigo carmine solution. If the selection criteria are met, randomization is performed and the formation is removed either by the ESD or EMR method.

EMR technique. 3-4 ml of a high-osmolar solution or saline solution stained with indigo carmine is injected into the submucosal layer under the formation. The formation is removed with the surrounding mucous membrane (at least 5 mm from the edge of the formation) using the standard diathermic polypectomy loop available to the operator. The formation is removed using electric current in the EndocatQ mode (ensuring alternating cutting and coagulation under the control of a processor built into the electrical unit). After removal of the formation, the resection site is examined in white light, then virtual chromoscopy (NBI), and then examination with magnification. The examination results are recorded in the scientific protocol separately, and are assessed as a whole. The criteria for visual removal of the formation within healthy tissues is the absence of visible fragments of the formation.

If residual tissue of the formation is detected, they are removed using the same technique. If the removal of residual tissue of the formation was performed by another method, indicate which one and why.

After the final assessment of the edges of the post-resection wound, 1 fragment is taken from each edge for morphological confirmation of R0 resection in the vertical edge (4 fragments in total) After EMR, in half of the cases (according to the instructions of the randomized recording), ablation of the edges with a polypectomy loop is performed.

The removed formation is extracted using a snare loop, if removed in parts, then all fragments, if possible, are extracted through the aspiration channel of the endoscope, for large fragments, a snare loop is used. A specimen not sent for morphological examination is considered lost.

ESD technique. After assessing the boundaries of the formation, a mark is made on it, retreating at least 5 mm from the edge, then a circular or semicircular incision of the mucosa will be made, after which the formation will be removed by dissection of the submucosal layer using a scarecrow knife, a knife with a ceramic head at the end in EndocutQ mode, spray-coag swift-coag. The ESD technique - tunnel method, where feasible, will also be used. The essence of the technique is a semilunar incision of the mucous membrane, retreating from the marks, and creating a tunnel under the formation to the proximal edge of the marks, with subsequent cutting off of the formation along the edges. The removed neoplasm is extracted and stretched on the plate. After removal, the edges and bottom of the wound are assessed, if necessary, prophylactic coagulation of visible vessels and clipping are performed.

Terminology (complications). Complications (adverse events) will be considered as occurring during the intervention (intraoperative), if they develop from the moment of insertion of the colonoscope until its removal. Otherwise, complications will be regarded as postoperative.

Perforation during the examination is diagnosed when the "target" symptom is detected - the presence of an additional ring-shaped structure at the bottom of the wound and/or during endoscopic visualization of a through defect in the organ wall.

Delayed perforation will be defined as the development of symptoms of peritoneal irritation and free gas in the abdominal cavity in the patient and/or the detection of a perforation hole in the area of removal of the formation during surgical revision.

Immediate (intraoperative) bleeding is bleeding that has not stopped within 4 minutes (the norm of hemostasis for capillary bleeding /from a finger/ according to Duke: onset after 2 minutes, end after 4 minutes) after removal of the formation and requiring one of the methods of endoscopic hemostasis (injection of adrenaline solution and/or coagulation (including ARS) and/or clipping.

Delayed bleeding is blood in the stool and unstable vital signs and/or a drop in hemoglobin ≥ 2 g / dl.

Postcoagulation syndrome is defined as the presence of abdominal pain and/or leukocytosis in the patient, an increase in C reactive protein and/or fever (more than 37.2) and/or symptoms of peritoneal irritation in the case of:

1. The absence of these symptoms before the manipulation and other reasons for their appearance
2. The absence of free gas in the abdominal cavity and/or detection perforation in the area of removal of the formation during surgical revision.

Methodology for morphological examination of preparations. After the preparation is removed in single fragments, it is fixed in a straightened state on a tight footrest. In the case of removal of the formation in fragments, the extracted fragments are also fixed in the above-mentioned manner, if possible. After fixation, the preparation is placed in a 10% formalin solution and delivered to the pathological anatomy department.

After 24 hours of fixation, the specimen is removed from formalin. Then the size of the formation is measured and parallel sections are made every 2-3 mm, which are placed in cassettes and undergo a standard procedure for preparing paraffin blocks, after which paraffin sections are made every 3-4 μm and a routine procedure for staining with hematoxylin and eosin. During the histological description of the specimen, it is planned to note the following parameters: number of fragments; size of the formation; its morphological type and differentiation; presence of a muscular plate of the mucosa, presence and thickness of submucosal tissue, diameter of the largest vessel in the sample; presence of formation tissues along the horizontal and vertical boundaries of the formation.

R0 is understood as the absence of formation cells along the border (vertical and horizontal) of the coagulation line The morphological classification of the formation will be carried out according to the WHO classification and the Vienna classification (see Appendix). When evaluating biopsies from the edges of the wound, the presence/absence of residual tissue of the formation (adenoma and/or adenocarcinoma and/or serrated formation) in the biopsy is indicated.

Documentation and computer statistical data processing. A separate medical record will be filled out for each patient in a closed database on the Internet.

Required - endophotographs of the formation before its removal and the wound after the end of the intervention, allowing to evaluate the parameters included in the analysis.

Statistical processing of the obtained data will be performed by the method of variation statistics with the calculation of the arithmetic mean, standard deviation, standard error of the mean and the reliability criterion (p). Differences at a significance level of 95% at p<0.05 are considered reliable. In order to check the significance of the difference between the means in different groups by comparing the variances of these groups, it is planned to use the methods of ANOVA (from the English ANalysis Of VAriance) analysis of variance. The Pearson correlation coefficient will be calculated to assess the presence or absence of a linear relationship between two variables and the tightness of this relationship. Calculations are planned to be made using the statistical section of the Microsoft Office Excel spreadsheet software package.

ELIGIBILITY:
Inclusion Criteria:

* Patient with benign non-invasive epithelial formations of the colon on a broad base (Is and II types), 20-60 mm in size
* Age ≥ 18 years.
* Signed informed voluntary consent for colonoscopy and removal of formations using the studied methods of EMR and ESD

Exclusion Criteria:

* . More than one large epithelial lesion on a broad base
* Colon lesion less than 20 mm and more than 60 mm
* Recurrent lesion.
* Reasonable suspicion of an invasive lesion (cancer), including one with submucosal invasion based on the results of preoperative assessment (NICE - 3; JNET - 3; Kudo - Vn).
* Presence of widespread malignant tumour in any part of the colon.
* Use of other methods of endoscopic lesion removal.
* IBD.
* Infectious disease requiring systemic therapy
* Patient on haemodialysis
* Uncorrectable coagulopathy (INR> 1.5), inability to discontinue antithrombotic drugs.
* Refusal to participate in the study. 12. General contraindications to endoscopic examination.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Radicality of removal | 1 months after removal
  Based on the pathomorphological report, the radicality of the removal of the epithelial formation by the EMR and ESD methods will be assessed. (R0, R1, Rx)
Duration of the operation | at the time of the operation
  from the moment of submucosal injection until the complete removal of the formation, the duration of the operation will be recorded
Intraoperative complications | at the time of the operation
  During the operation, intraoperative complications that arise are recorded: perforation, bleeding.
Postoperative complications | 1 months after removal
  Postoperative complications that arise from 1 day to 30 days after removal are assessed: postcoagulation syndrome, bleeding, perforation.
Relapse of education | 6 and 12 months after removal
  The postoperative scar is assessed for the presence of recurrent formation

SECONDARY OUTCOMES:
Endoscopic evaluation of submucous fibrosis | at the time of the operation
  During the operation, the degree of submucous fibrosis F0/F1/F2 is assessed according to the endoscopic classification.

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Gorbachev, Study Chair — Pirogov Russian National Research Medical University
Locations (1):
- Evgeny Gorbachev, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No